CLINICAL TRIAL: NCT07369310
Title: Randomized Trial on DBS Programming Based on Biomarkers vs. Standard Monopolar Review
Brief Title: Comparing Biomarker-Guided DBS Programming With Standard Clinical Monopolar Programming
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Ignacio Aracil Bolanos, MD PhD, Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIBSP-PTA-2024-62
Record Dates: First submitted 2026-01-21; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Parkinson's Disease; Parkinson; Parkinsons Disease (PD); Motor Fluctuations; DBS; Deep Brain Stimulation
Keywords: Parkinson's Disease; Deep Brain Stimulation; DBS Programming; Monopolar Review; Local Field Potentials; Beta Oscillations; BrainSense; Medtronic Percept; Neuroimaging-Guided Programming; Objective Programming; Adaptive Deep Brain Stimulatoin; Wearable Sensors; Inertial Sensors; Motor Fluctuations; OFF Time; Dyskinesia; Neuromodulation; Subthalamic Nucleus
MeSH Terms: conditions — Parkinson Disease; Dyskinesias | interventions — Diagnostic Imaging

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Conventional DBS Programming (Monopolar Review) (Active Comparator): Participants in this arm will undergo DBS programming using the conventional clinical approach based on monopolar review.
  Interventions: Device: Conventional DBS Programming (Monopolar Review)
- Objective-Guided DBS Programming (Imaging + Local Field Potentials) (Experimental): Participants in this arm will undergo DBS programming guided by objective markers. Selection of stimulation contacts will be informed by postoperative anatomical reconstruction of electrode location using Brainlab Elements™ and by beta-band local field potential (LFP) activity recorded with BrainSense™ from the implanted DBS system.
  Interventions: Device: Objective-Guided DBS Programming (Imaging and Local Field Potential-Based)

INTERVENTIONS:
Device: Conventional DBS Programming (Monopolar Review) — DBS programming performed using the conventional clinical monopolar review approach. Stimulation contacts and parameters are selected through systematic clinical testing based on clinician assessment of motor benefit and stimulation-related side effects, together with patient-reported symptoms. Programming does not incorporate postoperative electrode localization from neuroimaging or neurophysiological biomarkers. All participants are implanted with a CE-marked DBS system (Percept™ PC or RC with SenSight™ leads), and programming begins approximately 5 weeks after surgery following standard clinical practice.
  At 3 months after initial programming, Adaptive DBS is activated in all patients.
  Arms: Conventional DBS Programming (Monopolar Review)
Device: Objective-Guided DBS Programming (Imaging and Local Field Potential-Based) — DBS programming guided by objective anatomical and neurophysiological markers. Stimulation contact selection is informed by postoperative electrode reconstruction using Brainlab Elements™ and by LFP activity recorded with BrainSense™ from the implanted DBS system. These objective data are integrated with standard clinical testing to guide programming decisions. All participants are implanted with the same CE-marked DBS system (Percept™ PC or RC with SenSight™ leads), and programming starts approximately 5 weeks after surgery, following the same schedule as the comparator arm.
  At 3 months after initial programming, Adaptive DBS will be activated in all patients.
  Arms: Objective-Guided DBS Programming (Imaging + Local Field Potentials)

SUMMARY:
The goal of this clinical trial is to learn whether an objective, data-guided approach to programming deep brain stimulation (DBS) can improve motor outcomes in people with Parkinson's disease who undergo DBS surgery. The study includes adults aged 30 to 70 years with Parkinson's disease who are candidates for DBS.

The main questions it aims to answer are:

Does DBS programming based on objective markers (brain imaging and brain signals) reduce the amount of daily time patients spend in the OFF state more than conventional clinical programming?

Does this programming approach improve quality of life and motor symptoms compared with standard programming?

Researchers will compare conventional DBS programming based on clinical monopolar review with DBS programming guided by electrode location on neuroimaging and beta brain signals recorded from the implanted device, to see if the objective approach leads to better motor control and less OFF time.

Participants will:

Undergo DBS surgery using a clinically approved DBS system

Be randomly assigned to one of two DBS programming strategies

Wear inertial sensors at home for several days at different time points to objectively measure motor symptoms

Attend scheduled clinical visits for DBS programming and motor and non-motor assessments

Have adaptive DBS activated after 3 months and continue follow-up until 6 months after programming begins

DETAILED DESCRIPTION:
Deep brain stimulation (DBS) is an established therapy for patients with Parkinson's disease (PD) with motor fluctuations inadequately controlled by medication. However, DBS programming is currently based on monopolar review, a time-consuming process that relies heavily on clinician experience and subjective patient feedback. This approach does not systematically incorporate objective anatomical or neurophysiological information regarding the optimal stimulation contact and may require several months to achieve satisfactory clinical benefit.

Recent advances in DBS technology allow the integration of objective markers into the programming process. These include postoperative anatomical reconstruction of electrode location using neuroimaging and the recording of local field potentials (LFPs), particularly beta-band activity, from implanted DBS systems. In parallel, wearable inertial sensors enable continuous, objective quantification of motor states such as OFF time, dyskinesias, motor fluctuations, and gait disturbances in daily life.

This study is a pilot, randomized, controlled, parallel-group clinical trial with single-blind assessment, designed to evaluate whether DBS programming guided by objective markers (electrode localization on neuroimaging combined with beta LFP sensing) improves clinical outcomes compared with conventional programming based on monopolar clinical review. The study will be conducted in patients with Parkinson's disease undergoing DBS surgery at the Movement Disorders Unit of the Hospital de la Santa Creu i Sant Pau.

A total of 20 participants with idiopathic Parkinson's disease will be enrolled and randomized in a 1:1 ratio to one of two programming strategies: (1) conventional DBS programming based on clinical monopolar review, or (2) DBS programming guided by anatomical electrode reconstruction using Brainlab Elements™ and neurophysiological beta biomarkers obtained via BrainSense™. All participants will be implanted with a clinically approved DBS system (Percept™ PC or RC with SenSight™ directional leads, Medtronic) and will wear PDMonitor® inertial sensors for objective motor assessment. The only difference between groups is the DBS programming strategy.

All participants will undergo a 7-day PDMonitor® recording and a full clinical evaluation during the preoperative visit. DBS surgery will be followed by an approximately one-month postoperative period without stimulation. Initial DBS programming will begin around week 5 after surgery. A mid-programming clinical evaluation and PDMonitor® recording will be performed at approximately week 9. At 3 months after initiation of programming, participants will complete another 7-day PDMonitor® recording and a full clinical assessment, which will serve as the primary endpoint evaluation. Adaptive DBS (aDBS) will then be activated in both groups. A final follow-up visit at 6 months will include clinical assessments and sensor-based measurements; these post-aDBS data will be analyzed descriptively and exploratorily only.

The primary outcome is the percentage change in daily time spent in the OFF state between baseline (preoperative PDMonitor® recording) and 3 months after the start of DBS programming. Secondary outcomes include changes in quality of life measured by the PDQ-39, motor symptoms and motor complications assessed by the MDS-UPDRS parts III and IV, and non-motor symptoms assessed by the MDS-NMS, all between baseline and 3 months. Exploratory outcomes include descriptive changes in motor and functional measures between months 3 and 6 after activation of adaptive DBS.

PDMonitor® is used exclusively as a research assessment tool and does not constitute a therapeutic intervention. All implanted DBS devices, imaging reconstruction tools, and adaptive stimulation algorithms are CE-marked and used within their approved clinical indications.

The statistical analysis will follow a Bayesian framework appropriate for a pilot randomized study. Descriptive analyses will be performed for all variables. Bayesian linear mixed-effects models will be used to compare changes from baseline to 3 months between groups for the primary and secondary outcomes. Results will be expressed using posterior distributions, 95% credible intervals, Bayes factors, and comparison with a region of practical equivalence (ROPE). Analyses will be conducted primarily on an intention-to-treat basis, with per-protocol and sensitivity analyses to assess robustness. Missing data will be handled using Bayesian or multiple imputation methods as appropriate, except for the primary outcome, which will not be imputed in the absence of valid PDMonitor® recordings.

The study is exploratory in nature and is not designed as a confirmatory efficacy trial. It will be conducted in accordance with Good Clinical Practice (ICH-E6), the Declaration of Helsinki, and applicable European and Spanish data protection regulations. All participants will provide written informed consent prior to inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Age between 30 and 70 years.
* Confirmed diagnosis of idiopathic Parkinson's disease according to the MDS diagnostic criteria (Postuma et al., 2015).
* Indication for deep brain stimulation surgery based on CAPSIT-PD criteria.

Exclusion Criteria:

* Presence of severe surgical complications (e.g., intracranial hemorrhage, infection).
* Postoperative adverse events requiring electrode repositioning.
* Any other medical or neurological condition that could interfere with safe participation in the trial.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Daily OFF Time Assessed by Wearable Sensors | From baseline (preoperative 7-day recording) to 3 months after start of DBS programming
  Percentage change in daily time spent in the OFF state, measured objectively using PDMonitor® inertial sensors. OFF time will be quantified from continuous 7-day recordings performed at baseline (preoperative) and at 3 months after initiation of DBS programming. The outcome reflects motor fluctuations in real-life conditions.

SECONDARY OUTCOMES:
Change in Quality of Life (PDQ-39 Total Score) | From baseline to 3 months after start of DBS programming
  Change in health-related quality of life assessed using the Parkinson's Disease Questionnaire-39 (PDQ-39). The total score and domain scores will be compared between baseline and 3 months after initiation of DBS programming to evaluate the impact of programming strategy on patient-reported outcomes.
Change in Motor Symptoms (MDS-UPDRS Part III) | From baseline to 3 months after start of DBS programming
  Change in motor symptom severity assessed by the Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS), Part III. Scores obtained at baseline and at 3 months after initiation of DBS programming will be compared between groups.
Change in fluctuation severity (MDS-UPDRS Part IV) | From baseline and at 3 months after initiation of DBS programming.
  Changes in fluctuation severity assessed by the Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS), Part IV. Scores obtained at baseline and at 3 months after initiation of DBS programming will be compared between groups.
Change in Non-Motor Symptoms (MDS-NMS) | From baseline to 3 months after start of DBS programming
  Change in non-motor symptom burden assessed using the Movement Disorder Society Non-Motor Symptoms Scale (MDS-NMS). Total scores will be compared between baseline and 3 months after initiation of DBS programming.

OTHER OUTCOMES:
Effect of Adaptive DBS on Daily OFF Time Assessed by Wearable Sensors | From 3 months to 6 months after start of DBS programming
  Change in daily time spent in the OFF state assessed by PDMonitor® inertial sensors following activation of adaptive deep brain stimulation (aDBS). OFF time will be quantified from continuous 7-day recordings performed at 3 months after baseline (prior to initiation of aDBS programming) and at 6 months after baseline.
  Analyses are exploratory and descriptive. Between-group comparisons will also be performed as subgroup analyses according to assigned DBS programming strategy.
Effect of Adaptive DBS on Quality of Life (PDQ-39 Total Score) | From 3 months to 6 months after start of DBS programming
  Change in health-related quality of life assessed by the Parkinson's Disease Questionnaire-39 (PDQ-39) following activation of adaptive deep brain stimulation (aDBS). Total PDQ-39 scores obtained at 3 months after baseline (prior to initiation of aDBS programming) and at 6 months after baseline will be compared.
  Analyses are exploratory and descriptive. Between-group comparisons will also be performed as subgroup analyses according to assigned DBS programming strategy.
Effect of Adaptive DBS on Motor Symptoms (MDS-UPDRS Part III) | From 3 months to 6 months after start of DBS programming
  Descriptive evaluation of changes in motor symptom severity following activation of adaptive deep brain stimulation (aDBS), assessed using the Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS), Part III. Scores obtained at 3 months after baseline (prior to initiation of aDBS programming) and at 6 months after baseline will be compared.
  Analyses are exploratory and descriptive. Between-group comparisons will also be carried out as subgroup analyses according to assigned DBS programming strategy.
Effect of Adaptive DBS on Motor Fluctuations (MDS-UPDRS Part IV) | From 3 months to 6 months after start of DBS programming
  Descriptive evaluation of changes in motor fluctuation severity following activation of adaptive deep brain stimulation (aDBS), assessed using the Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS), Part IV. Scores obtained at 3 months after baseline (prior to initiation of aDBS programming) and at 6 months after baseline will be compared.
  Analyses are exploratory and descriptive. Between-group comparisons will also be carried out as subgroup analyses according to assigned DBS programming strategy.
Effect of Adaptive DBS on Non-Motor Symptoms (MDS-NMS) | From 3 months to 6 months after start of DBS programming
  Descriptive evaluation of changes in non-motor symptom burden following activation of adaptive deep brain stimulation (aDBS), assessed using the Movement Disorder Society Non-Motor Symptoms Scale (MDS-NMS). Total scores will be compared between assessments performed at 3 months after baseline (prior to initiation of aDBS programming) and at 6 months after baseline.
  Analyses are exploratory and descriptive. Between-group comparisons will also be carried out as subgroup analyses.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made publicly available. De-identified data may be shared upon reasonable request with the study investigators, subject to approval of a methodologically sound proposal, institutional review board approval as applicable, and execution of a data use agreement.

REFERENCES:
- [Background] Muller M, van Leeuwen MFC, Hoffmann CF, van der Gaag NA, Zutt R, van der Gaag S, Schouten AC, Contarino MF. From subthalamic local field potentials to the selection of chronic deep brain stimulation contacts in Parkinson's disease - A systematic review. Brain Stimul. 2025 Sep-Oct;18(5):1499-1510. doi: 10.1016/j.brs.2025.08.004. Epub 2025 Aug 11. PMID 40803531
- [Background] Neumann WJ, Gilron R, Little S, Tinkhauser G. Adaptive Deep Brain Stimulation: From Experimental Evidence Toward Practical Implementation. Mov Disord. 2023 Jun;38(6):937-948. doi: 10.1002/mds.29415. Epub 2023 May 6. PMID 37148553
- [Background] Shah A, Nguyen TK, Peterman K, Khawaldeh S, Debove I, Shah SA, Torrecillos F, Tan H, Pogosyan A, Lachenmayer ML, Michelis J, Brown P, Pollo C, Krack P, Nowacki A, Tinkhauser G. Combining Multimodal Biomarkers to Guide Deep Brain Stimulation Programming in Parkinson Disease. Neuromodulation. 2023 Feb;26(2):320-332. doi: 10.1016/j.neurom.2022.01.017. Epub 2022 Feb 24. PMID 35219571